CLINICAL TRIAL: NCT06086834
Title: Comparative Effects of McKenzie Retraction and Bruegger's Exercises on Forward Head Posture Among Young Adults
Brief Title: McKenzie Retraction and Bruegger's Exercises Effects on Forward Head Posture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0158
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Forward Head Posture
Keywords: Bruegger's Exercise; Forward head posture; McKenzie Exercise; Young Adult

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McKenzie Retraction Exercises (Experimental): McKenzie Retraction Exercises along with hot pack.
  Interventions: Other: McKenzie Retraction Exercises
- Bruegger's Exercise (Experimental): Bruegger's Exercise along with hot pack.
  Interventions: Other: Bruegger's Exercise

INTERVENTIONS:
Other: McKenzie Retraction Exercises — McKenzie Retraction exercises 5 days a week and 10-15 times for active exercises and 5-6 repetitions of clinician assisted exercise for a period of 4 weeks and a rest interval of 2 minutes between exercises.
  Arms: McKenzie Retraction Exercises
Other: Bruegger's Exercise — Bruegger's Exercise will be started from 10 seconds hold to 30 seconds with 2 seconds increment in every session. Rest time will be 30 seconds, 4 sets 12 times repetition, for duration of 30 mins per session, 5 days a week for a period of 4 weeks.
  Arms: Bruegger's Exercise

SUMMARY:
The aim of the study is to compare effects of McKenzie Retraction exercises and Bruegger's exercise on neck pain, ROM, craniovertebral angle and functional performance on forward head posture among young adults.

DETAILED DESCRIPTION:
There are many advantages of technology such as improving work productivity and efficacy; however, using technology for an extended period of time can place a substantial amount of load on the neck musculature leading to musculoskeletal disorder. The most related cause of neck pain is muscle weakness leading to forward head posture due to static abnormal posture used while using electronic devices.

The aim of the study is to compare effects of McKenzie Retraction exercises and Bruegger's exercise on neck pain, ROM, craniovertebral angle and functional performance on forward head posture among young adults. A randomized clinical trial will be conducted at Sadiq Hospital, Sargodha. Non-probability convenience sampling will be used, and 36 subjects, age 15-30 years will be randomly allocated into two groups by lottery method after meeting the inclusion criteria. Both groups will receive hot pack for 10-15 minutes, as common treatment. Group A will be treated with McKenzie Retraction Exercises and Group B will be treated with Bruegger's Exercise.5 sessions per week and total20sessions for 4 weeks. The outcome measures will be conducted through NPRS, NDI, photogrammetry and goniometry before and after 4 weeks. Data will be analyzed using SPSS software version 26.

ELIGIBILITY:
Inclusion Criteria:

* Both Male and Female age between 15-30 years.
* Craniovertebral angle < 50.
* Electronic gadgets >6 hours a day.
* Neck pain from the previous 3 months.
* NPRS >3.
* NDI > 10.

Exclusion Criteria:

* Neck surgery or trauma.
* Torticollis.
* Subjects with diagnosed cases of discogenic disease.
* Subjects with migraine problem.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 4th week.
  Changes from Baseline Numeric Pain Rating Scale (NRS-11), which is an eleven-point scale in which the end points are the extremes of no pain at all (score of 0) and the worst pain the patient has ever experienced (score of 10). NPRS-11 pain severity score of "4" is frequently given special significance in this regard, suggesting it as a potential threshold value for pain severity in clinical practice.
  This scale has high reliability (0.95-0.96).
NECK DISABILITY INDEX (NDI) | 4th week
  Changes from Baseline, In 1991, Howard Vernon developed the Neck Disability Index (NDI).The Neck Disability Index (NDI) was the first tool to measure self-reported disability in patients with neck pain. It is used extensively in literature and its psychometric properties have been well established. It has been translated and cross-culturally adapted to many languages. The index has 10 neck-related functional activities scored on a 0-5 scale for each item and a total raw score of 50. The higher the score, the greater the disability.
PHOTOGRAMMETRY | 4th week
  Changes from Baseline, The CVA was assessed using a digital camera. The camera was placed 1.5 m away from the participant's right side to take a lateral photographic view of the participant's head and neck in a seated position. The CVA is the angle between the horizontal line passing the 7th Cervical vertebra (C7) and then the line extending from C7 to the tragus of the ear. The resulting FHP was determined using Image J software. A CVA of less than 50º was defined as FHP. 'Image J', an analysis software with high reliability and validity.
UNIVERSAL GONIOMETER (ROM Cervical Spine Flexion) | 4th week
  Changes from Baseline ROM range of motion of cervical spine flexion was taken with help of goniometer. Goniometry, the measurement of joint angles, traditionally performed with a universal goniometer (UG), is a commonly utilized assessment tool in monitoring problems of the musculoskeletal system, as well as the progression of rehabilitation interventions.
UNIVERSAL GONIOMETER (ROM Cervical Spine Extension) | 4th week
  Changes from Baseline ROM range of motion of cervical spine flexion was taken with help of goniometer. Goniometry, the measurement of joint angles, traditionally performed with a universal goniometer (UG), is a commonly utilized assessment tool in monitoring problems of the musculoskeletal system, as well as the progression of rehabilitation interventions.
UNIVERSAL GONIOMETER (ROM Cervical Spine rotation) | 4th week
  Changes from Baseline ROM range of motion of cervical spine flexion was taken with help of goniometer. Goniometry, the measurement of joint angles, traditionally performed with a universal goniometer (UG), is a commonly utilized assessment tool in monitoring problems of the musculoskeletal system, as well as the progression of rehabilitation interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Amjad, MPhil, Principal Investigator — Riphah International University
Locations (1):
- Sadiq Hospital, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heydari Z, Sheikhhoseini R, Shahrbanian S, Piri H. Establishing minimal clinically important difference for effectiveness of corrective exercises on craniovertebral and shoulder angles among students with forward head posture: a clinical trial study. BMC Pediatr. 2022 Apr 27;22(1):230. doi: 10.1186/s12887-022-03300-7. PMID 35477430
- [Background] Sarraf F, Varmazyar S. Comparing the effect of the posture of using smartphones on head and neck angles among college students. Ergonomics. 2022 Dec;65(12):1631-1638. doi: 10.1080/00140139.2022.2047229. Epub 2022 May 4. PMID 35199629
- [Background] Suwaidi ASA, Moustafa IM, Kim M, Oakley PA, Harrison DE. A Comparison of Two Forward Head Posture Corrective Approaches in Elderly with Chronic Non-Specific Neck Pain: A Randomized Controlled Study. J Clin Med. 2023 Jan 9;12(2):542. doi: 10.3390/jcm12020542. PMID 36675471
- [Background] Augustsson SR, Reinodt S, Sunesson E, Haglund E. Short-term effects of postural taping on pain and forward head posture: a randomized controlled trial. BMC Musculoskelet Disord. 2022 Feb 19;23(1):162. doi: 10.1186/s12891-022-05083-5. PMID 35183157
- [Background] Alvarez-Rodriguez J, Leiros-Rodriguez R, Morera-Balaguer J, Marques-Sanchez P, Rodriguez-Nogueira O. The Influence of the Locus of Control Construct on the Efficacy of Physiotherapy Treatments in Patients with Chronic Pain: A Systematic Review. J Pers Med. 2022 Feb 7;12(2):232. doi: 10.3390/jpm12020232. PMID 35207720
- [Background] Sterling M, de Zoete RMJ, Coppieters I, Farrell SF. Best Evidence Rehabilitation for Chronic Pain Part 4: Neck Pain. J Clin Med. 2019 Aug 15;8(8):1219. doi: 10.3390/jcm8081219. PMID 31443149
- [Background] Takasaki H, Yamasaki C. Immediate neck hypoalgesic effects of craniocervical flexion exercises and cervical retraction exercises among individuals with non-acute neck pain and a directional preference for retraction or extension: preliminary pretest-posttest randomized experimental design. J Man Manip Ther. 2023 Oct;31(5):368-375. doi: 10.1080/10669817.2023.2201918. Epub 2023 Apr 13. PMID 37052492
- [Background] Abdel-Aziem AA, Mohamed RR, Draz AH, Azab AR, Hegazy FA, Diab RH. The effect of McKenzie protocol vs. deep neck flexor and scapulothoracic exercises in subjects with chronic neck pain - a randomized controlled study. Eur Rev Med Pharmacol Sci. 2022 May;26(9):3138-3150. doi: 10.26355/eurrev_202205_28731. PMID 35587064
- [Background] Kim DH, Kim CJ, Son SM. Neck Pain in Adults with Forward Head Posture: Effects of Craniovertebral Angle and Cervical Range of Motion. Osong Public Health Res Perspect. 2018 Dec;9(6):309-313. doi: 10.24171/j.phrp.2018.9.6.04. PMID 30584494
- [Background] Al-Hadidi F, Bsisu I, AlRyalat SA, Al-Zu'bi B, Bsisu R, Hamdan M, Kanaan T, Yasin M, Samarah O. Association between mobile phone use and neck pain in university students: A cross-sectional study using numeric rating scale for evaluation of neck pain. PLoS One. 2019 May 20;14(5):e0217231. doi: 10.1371/journal.pone.0217231. eCollection 2019. PMID 31107910
- [Background] Perez-de la Cruz S, de Leon OA, Mallada NP, Rodriguez AV. Validity and intra-examiner reliability of the Hawk goniometer versus the universal goniometer for the measurement of range of motion of the glenohumeral joint. Med Eng Phys. 2021 Mar;89:7-11. doi: 10.1016/j.medengphy.2021.01.005. Epub 2021 Jan 27. PMID 33608127
- [Background] Bergh A, Lauridsen NG, Hesbach AL. Concurrent Validity of Equine Joint Range of Motion Measurement: A Novel Digital Goniometer versus Universal Goniometer. Animals (Basel). 2020 Dec 19;10(12):2436. doi: 10.3390/ani10122436. PMID 33352686
- [Background] Langenfeld A, Gassner AP, Wirth B, Muhlemann MB, Nyiro L, Bastiaenen C, Swanenburg J. Responsiveness of the German version of the Neck Disability Index in chronic neck pain patients: a prospective cohort study with a seven-week follow-up. Arch Physiother. 2022 Oct 17;12(1):23. doi: 10.1186/s40945-022-00149-y. PMID 36244985
- [Background] Farooq MN, Mohseni-Bandpei MA, Gilani SA, Hafeez A. Urdu version of the neck disability index: a reliability and validity study. BMC Musculoskelet Disord. 2017 Apr 8;18(1):149. doi: 10.1186/s12891-017-1469-5. PMID 28388888